CLINICAL TRIAL: NCT05150353
Title: Detection of Amyloid Deposits in the Wrist by MRI With Mapping and High Resolution Sequences in Systemic Amyloidosis
Brief Title: Detection of Amyloid Deposits in the Wrist by MRI With Mapping and High Resolution Sequences in Systemic Amyloidosis (AMYLOCARP)
Acronym: AMYLOCARP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2018-A00881-54 Promoteur
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Amyloid; Systemic Amyloidosis
MeSH Terms: conditions — Alzheimer Disease; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with cardiac amyloidosis (Experimental)
  Interventions: Procedure: MRI
- Healthy volunteers (Placebo Comparator)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Wrist MRI

SUMMARY:
This study is based on the hypothesis that MRI could make it possible to non-invasively detect these amyloid deposits at the level of the wrist using parametric sequences known as T1 mapping, in the form of an extension of T1 in the wrists. areas where amyloid deposits are found in the wrist.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Woman or man over 18 years old
* With ATTR or AL cardiac amyloidosis with or without carpal tunnel. The diagnosis of amyloidosis must be proven by a positive myocardial biopsy or diphosphonate scintigraphy.
* Affiliate or beneficiarie of a social security scheme.
* Having signed the free and informed consent.

Healthy volunteers:

* Woman or man over 18 years old
* Affiliate or beneficiarie of a social security scheme.
* Having signed the free and informed consent.

Exclusion Criteria:

Patient group:

* Patients participating in another clinical study.
* Patients suffering from rheumatoid arthritis or other autoimmune disease (vasculitis, lupus, scleroderma, etc.)
* Patients with a medical history of wrist surgery (exclude the operated side).
* Patients with a contraindication to performing an MRI (pacemaker, etc.)
* Pregnant or breastfeeding women.
* Protected patients: Adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision.

Healthy volunteer:

* Volunteers participating in another clinical study.
* Volunteers suffering from rheumatoid arthritis or other autoimmune disease (vasculitis, lupus, scleroderma, etc.)
* Pregnant or breastfeeding women.
* Volunteer with a contraindication to performing an MRI (pacemaker, etc.)
* Protected volunteers: Adults under guardianship, guardianship or other legal protection, deprived of their liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2022-04-24 (Estimated)

PRIMARY OUTCOMES:
T1 measurement (ms) associated with each of the 5 regions of interest at the wrist | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Paul d'Egine, Champigny-sur-Marne, France